CLINICAL TRIAL: NCT02662816
Title: Feasibility Study of the Quantification of Glutathione Concentrations in Muscle and Liver Using in Vivo Proton Magnetic Resonance Spectroscopy (1H MRS)in Human
Brief Title: Non-invasive Quantification of Muscle and Liver Glutathione GSH-MRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: UMR 1019 Unité de Nutrition Humaine (Unknown); Laboratoire Régional de Nutrition Humaine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-0253; 2015-A01426-43 (Registry Identifier: 2015-A1426-43)
Record Dates: First submitted 2015-12-22; First posted 2016-01-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Assay Muscle; Liver Glutathione in Healthy Human
Keywords: Glutathione; Liver; Muscle; Proton magnetic resonance spectroscopy; Healthy human
MeSH Terms: interventions — Proton Magnetic Resonance Spectroscopy

ARMS (1):
- glutathion (Experimental): The study will validate the detection and the quantification of glutathione in muscle and liver using 1H MRS
  Interventions: Device: Proton magnetic resonance spectroscopy (1H MRS); Other: a protein rich breakfast at home; Other: a protein rich lunch at the Clinical Investigation Center

INTERVENTIONS:
Device: Proton magnetic resonance spectroscopy (1H MRS)
Other: a protein rich breakfast at home
Other: a protein rich lunch at the Clinical Investigation Center

SUMMARY:
Glutathione (glutamyl-cysteinyl-glycine) is the main intracellular compound. It participates also in the detoxification of electrophiles molecules of which paracetamol. It is synthesized in the liver during the postprandial phase, which establishes a stock that is mobilized for the other tissues (muscle)during the postabsorptive period. It is of common knowledge that the decrease in glutathione concentrations associated with ageing could be involved in the development of the degenerative pathologies linked to the old age. These changes could be reversed by an increase in dietary cysteine, the amino acid limiting of the endogenous synthesis of GSH. The development of nutritional strategies aiming at an improvement of the status glutathione requires the determination of its concentration within tissues, where it is active. The quantification of tissue concentrations of glutathione by biochemical techniques requires tissue biopsies. Such a method can be performed for the muscle, but liver biopsy is not feasible outside of a surgery. It is necessary to set up a non-invasive method to quantify muscle and liver glutathione.

DETAILED DESCRIPTION:
The study will validate the detection and the quantification of glutathione in muscle and liver using 1H MRS. The accuracy of the method will be assessed from intra and inter-volunteer measurements. 1H MRS measurements will be performed with the Magnetic Resonance Imaging (MRI) 3 Tesla system of the Hospital, twice for each volunteer.

Prior to the measurements, volunteers will have a protein rich breakfast at home and a protein rich lunch at the Clinical Investigation Center.

ELIGIBILITY:
Inclusion Criteria:

* - Healthy Volunteers, men or women, from 18 to 35 years old
* Having filled the questionnaire of compatibility in the MRI and having no contraindication in the MRI
* Having given their written, free and informed consent
* Affiliated with a social security system
* 19 < BMI < 25 kg.m-2

Exclusion Criteria:

* - Age < 18 ans ou > 35 ans
* BMI < 19 ou > 25 kg.m-2
* Carrier of a pacemaker, cochlear implants, metallic implants or magnetic element (cf questionnaire of compatibility in the MRI, Appendix 3)
* Under treatment with repeated doses of paracetamol during the 2 weeks preceding the inclusion
* Under treatment in N-acetylcysteine during 2 weeks preceding the inclusion
* Regular sporttraining > 3 hours / week
* Claustrophobia
* Difficulty of being immobile
* Pregnant women or women who are breast-feeding
* Incapacitated legal (private person of freedom or under guardianship)
* People who cannot be followed and/or compliant in the requirements of the study for psychological, social, family or geographical reasons,
* People already included in another clinical trial

Ages: 18 Days to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2016-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Signal-to-noise ratio of glutathione detected in liver and muscle | 2 h after the lunch.

SECONDARY OUTCOMES:
Glutathione concentrations in liver | 2 h after the lunch
Glutathione concentrations in muscle | 2 h after the lunch
Glutathione concentrations in means | 2 h after the lunch
Glutathione concentrations in intervariabilities | 2 h after the lunch
Glutathione concentrations in intravariabilities | 2 h after the lunch

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France